CLINICAL TRIAL: NCT00480701
Title: Evaluation of 123-I Iodobenzovesamicol (IBVM) and SPECT as a Marker of Acetylcholine Transporter Density in the Brain of Healthy Subjects and Patients With Alzheimer Disease
Brief Title: Evaluation of 123-I Iodobenzovesamicol (IBVM) and SPECT Imaging of Healthy Subjects and Patients With Alzheimer Disease
Acronym: IBVM001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IBVM001
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer Disease; Parkinson Disease
Keywords: Alzheimer; Parkinson; dementia; neurologic
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Dementia; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [123I]-IBVM (Experimental): To assess [123I] IBVM and SPECT imaging
  Interventions: Drug: [123I]-IBVM

INTERVENTIONS:
Drug: [123I]-IBVM — Subjects will be asked to undergo an injection of 123-I IBVM followed by up to three approximately thirty minute SPECT scans during the next 24 hours.

SUMMARY:
The underlying goal of this study is to assess 123-I IBVM SPECT imaging as a tool to assess cholinergic transporter binding in the brain of AD and PD research participants and age- and gender-matched healthy subjects.

DETAILED DESCRIPTION:
Approximately 25 patients with mild to moderate Alzheimer's disease (AD) and 25 patients Parkinson's disease and 20 healthy controls will be recruited to participate in this study.

AD patients will be eligible to participate if they have a diagnosis of AD based on NINCDS-ADRDA criteria.

PD patients will be eligible to participate if they have a clinical diagnosis of Parkinson's disease.

Healthy controls will be evaluated to ensure that there is no evidence of neurodegenerative changes including cognitive decline.

All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a physical and neurological evaluation and cognitive assessment.

Subjects will be asked to undergo an injection of 123-I IBVM followed by up to three approximately thirty minute SPECT scans during the next 24 hours.

Subjects may be asked to undergo a second imaging visit two-weeks to six months following the initial imaging visit to assess the reproducibility of the imaging outcome and/or the progressive change from baseline in 123-I IBVM binding.

The imaging analyses will be performed by an image-processing specialist who will remain masked to clinical diagnosis. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a target region to cerebellar ratio.

ELIGIBILITY:
Alzheimer's Inclusion Criteria:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Alzheimer's disease
* Mini-Mental Status Exam score >10 and < 25.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential or negative urine pregnancy test on day of 123-I IBVM injection.

Alzheimer's Exclusion Criteria:

* The subject has signs or symptoms of another neurodegenerative disease
* Subjects with an iodine allergy.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has received an investigational drug within 60 days before the screening visit.
* Pregnancy

Parkinson's Inclusion Criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Parkinson's disease
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential or negative urine pregnancy test on day of 123-I IBVM injection.

Parkinson's Exclusion Criteria:

* Subjects with an iodine allergy.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Does 123-I IBVM SPECT provide a quantitative measure of acetylcholinergic transporters in Healthy controls and AD patients? | 24 hours

SECONDARY OUTCOMES:
Does 123-I IBVM SPECT demonstrate reduced acetylcholinergic transporter binding in AD compared to healthy controls? | 1 year
Does 123-I IBVM SPECT provide a reliable measure of acetylcholinergic transporters in healthy controls and AD patients? | 2 weeks to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States